CLINICAL TRIAL: NCT01507519
Title: The First-In-Man Safety and Performance Evaluation of the Biomime Sirolimus Eluting Stent System for the Treatment of Patients With Single, De Novo, Non-Complex Coronary Lesions-The Biomime Pilot FiM Trial.
Brief Title: Study Safety and Performance of the Biomime Stent in Patients With Single, De Novo, Non-Complex Coronary Lesions
Acronym: meriT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Collaborators: Lifecare Institute of Medical Sciences and Research Ahmedabad Gujarat India (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOFIM/MLS/100209
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: BioMime™ Sirolimus-Eluting Coronary Stent System
Oversight: Data Monitoring Committee: No

ARMS (1):
- BioMime™ (Experimental): BioMime™ DES
  Interventions: Device: Sirolimus Eluting Coronary Stent System (Biomime)

INTERVENTIONS:
Device: Sirolimus Eluting Coronary Stent System (Biomime) — Coronary Artey PTCA
  Other Names: Biomime Sirolimus Eluting Stent System

SUMMARY:
1.) Indigenously developed and designed BioMimeTM is a

* predictably safe & efficacious 3rd generation drug eluting stent (DES)
* with a propensity to minimize vascular injury by use of an intelligent mix of ultra-low strut thickness Co-Cr stent,
* highly documented drug Sirolimus &
* a biocompatible, biodegradable polymer

DETAILED DESCRIPTION:
* Principal Investigator: Dr. Sameer Dani, Interventional Cardiologist, Life Care Hospital, Ahmedbad. Mobile +91 98250 38855.
* Study Title: The First-In-Man Safety and Performance Evaluation of the BiomimeTM Sirolimus-Eluting Stent System for the Treatment of Patients with Single, De novo, Non-complex Coronary Lesions - The BiomimeTM Pilot FiM Trial
* Sponsor: Meril Life Sciences Pvt. Ltd.
* Study device: BiomimeTM Sirolimus-Eluting Stent (BiomimeTM SES, Meril Life Sciences)
* Study objective: To evaluate the safety and efficacy of BiomimeTM SES.
* Study design: Phase IV, prospective study to be conducted in a single centre (Life Care Hospital, Ahmedbad)
* Study population: A total of 30 patients with stable or unstable coronary disease, or silent ischemia with documented evidence of ischemia, with angiography, and, in a pre-specified subset, intravascular ultrasound (IVUS) at 8-month follow-up.
* Participating Centre: Life Care Hospital, Ahmedabad
* QCA & IVUS core lab: To be decided.
* Follow-up: All patients will undergo clinical follow-up at 1, 6, 12 and 24 months. All patients will undergo angiographic follow-up at 8 months. All patients will be submitted to intravascular ultrasound at 8 months.
* Primary safety endpoint: Major Adverse Cardiac Events (MACE) at 30 days clinical follow-up. MACE defined as any of the following: cardiac death, myocardial infarction, and ischemia driven target lesion revascularization (TLR).
* Primary efficacy endpoint:
* In-stent luminal loss assessed by quantitative coronary angiography (QCA) at 8-month follow-up
* Percentage of in-stent volume obstruction measured by IVUS at 8- month follow-up.
* Secondary endpoints:
* Occurrence of Major Adverse Cardiac Events (MACE) defined as cardiac death, non-fatal acute myocardial infarction, and need for repeat target-lesion revascularization (by cardiac bypass graft or repeat percutaneous coronary intervention up to 24 months of follow-up.
* Angiographic binary restenosis at 8 months angiographic follow-up.
* Other endpoints:
* Rates of stent thrombosis (acute, sub-acute, late and very-late) up to 24 months follow-up
* In-stent and in-segment minimum lumen diameter (MLD) and % diameter stenosis (DS) by QCA at 8-month angiographic follow-up.
* In-stent acute gain by post procedure QCA.
* Late acquired incomplete stent apposition by IVUS at 8 month follow-up.
* Primary analysis: The primary endpoint will be analyzed for all subjects who had a de novo coronary lesion enrolled in this study (intention to treat)

ELIGIBILITY:
Inclusion Criteria:

* Patient with > 18 years of age;
* Symptoms of stable or unstable angina and/or presence of a positive functional test for ischemia;
* Presence of a single de novo target lesion located in a native coronary vessel suitable for percutaneous treatment with the study stents;
* Acceptable candidate for coronary artery bypass graft (CABG) surgery;
* The subject is willing to sign a written informed consent prior to procedure, and is willing to undergo ALL study protocol follow-ups, including angiographic (and IVUS) follow-ups at 8 months.

  * Target lesion located in a major epicardial coronary vessel with reference of 2.5-3.5mm in diameter (by visual estimation)
  * Target lesions ≤ 19mm in length (by visual estimation) that can be treated (covered) by one single study stent (19 or 24mm in length);
  * ≥ 50% and < 100% diameter stenosis;
  * TIMI (Thrombolysis In Myocardial Infarction) flow grade ≥ 2.

Exclusion Criteria:

* Known hypersensitivity or contraindication to mTOR inhibitor class drugs (sirolimus), heparin, any required medications including thienopyridines, cobalt chromium, and contrast media which cannot be adequately pre medicated;
* Patient is a female with childbearing potential;
* Pre-treatment of the target lesion with any devices other than balloon angioplasty;
* Previous brachytherapy in the target vessel;
* Presence of non-target vessel lesions which require staged procedure(s) < 30 days of the index procedure;
* Prior CABG surgery to target vessel;
* Previous percutaneous coronary intervention (PCI) or CABG surgery < 30 days to the index procedure date;
* Acute myocardial infarction < 3 days, with cardiac enzyme elevation including total creatine kinase (CK) > 2 times the upper normal limit value and/or CK-MB above the upper normal limit value within the past 72 hours;
* CK and/or CK-MB levels elevated above the upper normal limit value at the time of the index procedure;
* Documented left ventricular ejection fraction < 30%;
* Renal insufficiency determined by a baseline serum creatinine > 2.0/dl;
* Thrombocytopenia with a baseline platelet count < 100,000 cells/mm3;
* Anemia with baseline hemoglobin < 10g/dL;
* Extensive peripheral vascular disease or extreme anticoagulation that precludes safe > 5 French sheath insertion;
* History of bleeding diathesis, coagulopathy, or will refuse blood transfusions;
* Patients has suffered a stroke, transient ischemic attack (TIA), or cerebrovascular accident (CVA) within the past 6 months;
* Significant gastrointestinal or genitourinary bleed within the past 6 months;
* Patient is a recipient of a heart transplant;
* Any elective surgical procedure is planned within 12 months of the index procedure;
* Known illness or any serious clinical condition with life expectancy < 2 years;
* Participation in the active or follow-up phase of any other clinical trial within 6 months;
* Impossibility to comply with anti-platelet therapy during the study clinical follow-up;
* Any impossibility to comply with all protocol follow-ups.
* Target lesion or vessel with angiographic evidence of moderate or severe calcification;
* Presence of severe tortuosity;
* Presence of severe angulation (> 60o);
* Presence of intraluminal thrombus;
* Target lesion involving a bifurcation (side branch ≥ 2.0mm);
* Target lesion located in the left main stem;
* Aorto-ostial lesion location;
* Target lesion involving a side branch with reference diameter ≥ 2.0mm;
* Presence of a significant stenosis (> 40%) in the target vessel either proximal or distal to the target lesion that will be untreated;
* Previous placement of a stent within 10mm of the target lesion;
* Total occlusion (TIMI flow grade 0 or 1);
* Target lesion located in an arterial or vein graft;
* Target lesion due to in-stent restenosis;
* Coronary anatomy unsuitable for percutaneous treatment with implantation of the available study stents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
MACE at 30 days clinical F/U | 30 days
  Major Adverse Cardiac Events (MACE) at 30 days clinical follow-up. MACE defined as any of the following: cardiac death, myocardial infarction, and ischemia driven target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Angiographic Binary restenosis at 8-months F/U | 8-months post implant
  * Occurrence of Major Adverse Cardiac Events (MACE) defined as cardiac death, non-fatal acute myocardial infarction, and need for repeat target-lesion revascularization (by cardiac bypass graft or repeat percutaneous coronary intervention up to 24 months of follow-up.
  * Angiographic binary restenosis at 8 months angiographic follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: SAMEER DANI, MD;DM(Card.), Principal Investigator — Life Care Institute of Medical Sciences & Research Centre
Locations (1):
- Life Care Institute of Medical Sciences & Research, Ahmedabad, Gujarat, India

REFERENCES:
- See also: First in man study — https://www.ncbi.nlm.nih.gov/pubmed/23965355